CLINICAL TRIAL: NCT04626557
Title: Identifying Disease Mechanisms Underlying the Association Between Asthma and Infertility - The INFLammation Asthma Mechanism Endometrium (INFLAME) Study
Acronym: INFLAME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Casper Tidemandsen, MD, Hvidovre University Hospital
Other Study IDs: H-20029413
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Asthma; Infertility, Female
MeSH Terms: conditions — Asthma; Infertility, Female | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Endometrium biopsis
  * Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with astma: At the 7th -14th cycle day, an endometrium sample from the uterus lining will be obtained together with sputum, as indicators of the system inflammation expressed both in the lungs and the uterus, and blood samples.
  Interventions: Procedure: biopsy
- Women without asthma: At the 7th - 14th cycle day, an endometrium sample from the uterus lining will be obtained together with sputum, as indicators of the system inflammation expressed both in the lungs and the uterus, and blood samples.
  Interventions: Procedure: biopsy

INTERVENTIONS:
Procedure: biopsy — biopsy of the endometrium

SUMMARY:
To investigate if asthma affects the inflammatory balance of the endometrium and thereby interfere with implantation, as indicated by the characteristics of the inflammatory cells in the endometrium and airways in women with asthma who are referred for IUI or IVF due to infertility, compared to otherwise healthy women who are referred for IUI or IVF due to infertility.

DETAILED DESCRIPTION:
The link between asthma and fertility may be associated with widespread tissue inflammation, as inflammatory changes are not only affecting the respiratory organs, but also systemically, and here by affecting both the lungs and the reproductive organs in women with asthma.

A likely mechanism involved in infertility among asthmatic women seems to be inflammatory changes found in the endometrium of the uterus. Some studies show high number of mast cells, eosinophil granulocytes and basophil granulocytes in the endometrium[1]. One study found low values of VEGF in endometrial secretion in women with asthma as a possible cause for subfertility [2]. Others assume, that an imbalance of the adaptive immune system (both the Th1 and Th2/TH17 response) is associated with infertility [3].

It has been shown that inflammation in the endometrium with a specific combination of cytokines and chemokines is part of successful implantation [4]. However, If the inflammatory process is characterized by a less optimal combination of cytokines and chemokines the reproductive outcome may be less successful. The systemic inflammation caused by asthma could offset the balance between the cytokines and chemokines in the endometrium and thereby have negative impact on reproductive outcome.

In the present study, our aim is to analyze inflammation in the uterus and in the airways in women with asthma referred to fertility treatment receiving Intrauterine insemination (IUI) or in vitro fertilization (IVF) to characterize and thereby provide knowledge of the mechanisms underlying the association between asthma and reproductive outcomes.

In an explorative non-randomized study, including 30 participants divided into two groups: 15 women with asthma and 15 non-asthmatic controls. The patients will go through an asthma work-up (diagnosis, allergy, medication, and inflammation). Menstrual blood will be collected at home using the menstrual cup and at the 7th-14th day cycle day, an endometrium sample from the uterus lining will be obtained together with sputum, as indicators of the system inflammation expressed both in the lungs and the uterus, and blood samples.

ELIGIBILITY:
Inclusion criteria:

Asthma n= 15:

* Informed consent.
* Diagnosis of asthma.
* 18-40 years.
* Referred to Intra Uterine Insemination (IUI) or in vitro fertilization (IVF)

Non-asthmatic n= 15:

* Informed consent.
* 18-40 years.
* Referred to Intra Uterine Insemination (IUI) or in vitro fertilization (IVF)

Exclusion criteria:

Asthma only:

* Other respiratory diseases than asthma.
* Other inflammatory disease or a disease that affects fertility.
* Infections requiring antibiotics or anti-viral treatment within 30 days.
* Current smokers and/or life-time tobacco exposure > 10 pack-years.
* Endometriosis.
* Infertility due to other reasons than male factor, tubal factor or unexplained infertility.
* No pelvic inflammatory disease (PID) within the last 6 months.
* No contraceptive intrauterine device (IUD), or other contraceptive for the last 6 months.

Non-asthmatic controls:

* No respiratory diseases.
* Other inflammatory disease or a disease that affects fertility.
* Infections requiring antibiotics or anti-viral treatment within 30 days.
* Current smokers and/or life-time tobacco exposure > 10 pack-years.
* Endometriosis.
* Infertility due to other reasons than male factor, tubal factor or unexplained infertility.
* No pelvic inflammatory disease (PID) within the last 6 months.
* No contraceptive intrauterine device (IUD), or other contraceptive for the last 6 months.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: 30 participants divided into two groups: 15 women with asthma and 15 non-asthmatic controls. The patients will go through an asthma work-up (diagnosis, allergy, medication, and inflammation). Menstrual blood will be collected at home using the menstrual cup and at the 7th-14th cycle day, an endometrium sample from the uterus lining will be obtained together with sputum, as indicators of the system inflammation expressed both in the lungs and the uterus, and blood samples.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
type of inflammatory cells | 6 months
  To classify the type of inflammatory cells, (ie. cytokines and inflammatory cells), found in the uterine lining (endometrium) in women with asthma suffering from infertility, compared to non-asthmatic controls.

SECONDARY OUTCOMES:
airway inflammation vs inflammation in the endometrium. | 6 months
  Explore associations between airway inflammation and inflammation in the endometrium.
systemic inflammation vs local inflammation | 6 months
  Explore associations between systemic inflammation and local inflammation
Severity | 6 months
  Differences in local inflammation of the endometrium within different severities/phenotypes of asthma.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory Medicine, Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Will be shared upon request